CLINICAL TRIAL: NCT02649218
Title: An Open Label, Multicenter, Extension Study to Evaluate the Long-term Safety of QGE031 240 mg s.c. Given Every 4 Weeks for 52 Weeks in Chronic Spontaneous Urticaria Patients Who Completed Study CQGE031C2201
Brief Title: A Safety Extension Study to Evaluate the Long-term Safety of QGE031 in Chronic Spontaneous Urticaria (CSU) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQGE031C2201E1; 2015-003636-13 (EudraCT Number)
Record Dates: First submitted 2015-12-15; First posted 2016-01-07 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: QGE031; chronic; spontaneous; Urticaria; CSU; adults; Safety; ligelizumab
MeSH Terms: conditions — Chronic Urticaria; Bronchiolitis Obliterans Syndrome; Urticaria | interventions — ligelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ligelizumab (Experimental): QGE031 240 mg s.c. q4w x 13 treatments
  Interventions: Biological: Ligelizumab

INTERVENTIONS:
Biological: Ligelizumab — QGE031 240 mg s.c. q4w
  Other Names: QGE031

SUMMARY:
A safety extension study to evaluate the long-term safety of QGE031 240 mg s.c. given every 4 weeks for 52 weeks in Chronic Spontaneous Urticaria (CSU) patients who completed study CQGE031C2201

DETAILED DESCRIPTION:
A safety extension study to evaluate the long-term safety of QGE031 in Chronic Spontaneous Urticaria patients

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for inclusion in this study have to fulfill all of the following criteria:

  1. Written informed consent must be obtained before any assessment is performed.
  2. Patients who complete the treatment epoch in study CQGE031C2201 and complete at least Visit 203 (Week 32 of the follow-up epoch, ≥16 weeks after last injection) and present with active disease as defined by UAS7 ≥12.
  3. Patients must not have any missing eDiary entries in the 7 days prior to Visit 301 (patients are allowed to repeat until this criterion is met).
  4. Willing and able to complete a daily symptom eDiary for the duration of the study and adhere to the study visit schedules.

Exclusion Criteria:

Clearly defined underlying etiology for chronic urticaria other than chronic spontaneous urticaria

* Evidence of parasitic infection
* Any other skin diseases than chronic spontaneous urticaria with chronic itching
* Contraindications to or hypersensitivity to fexofenadine, loratadine, cetirizine, or epinephrine
* History of anaphylaxis
* History or current diagnosis of ECG abnormalities indicating significant risk of safety for patients participating in the study
* History of hypersensitivity to any of the study drugs or its components of similar chemical classes
* Pregnant or nursing (lactating) women Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (17):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Waldorf, Maryland
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Lake Oswego, Oregon
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, South Burlington, Vermont
- Australia (5):
  - Novartis Investigative Site, Campbelltown, New South Wales
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, East Melbourne, Victoria
- Canada (3):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Québec
- Germany (7):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Münster
- Greece (2):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Athens
- Japan (11):
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kamimashi-gun, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Saitama, Saitama
  - Novartis Investigative Site, Machida, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Shinagawa Ku, Tokyo
  - Novartis Investigative Site, Hiroshima
- Russia (4):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Smolensk
- Spain (9):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Alcorcón, Madrid
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Taiwan (3):
  - Novartis Investigative Site, Taoyuan District, Taiwan
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Novartis Investigative Site, Yeovil, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Metz M, Bernstein JA, Gimenez-Arnau AM, Hide M, Maurer M, Sitz K, Soong W, Sussman G, Hua E, Barve A, Barbier N, Balp MM, Severin T. Ligelizumab improves angioedema, disease severity and quality-of-life in patients with chronic spontaneous urticaria. World Allergy Organ J. 2022 Nov 15;15(11):100716. doi: 10.1016/j.waojou.2022.100716. eCollection 2022 Nov. PMID 36440464
- [Derived] Maurer M, Gimenez-Arnau A, Bernstein JA, Chu CY, Danilycheva I, Hide M, Makris M, Metz M, Savic S, Sitz K, Soong W, Staubach P, Sussman G, Barve A, Burciu A, Hua E, Janocha R, Severin T. Sustained safety and efficacy of ligelizumab in patients with chronic spontaneous urticaria: A one-year extension study. Allergy. 2022 Jul;77(7):2175-2184. doi: 10.1111/all.15175. Epub 2021 Nov 22. PMID 34773261
- See also: Core study — https://clinicaltrials.gov/ct2/show/NCT02477332?term=cqge031c2201&draw=2&rank=2
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the subjects who completed core study (NCT02477332) that were eligible for extension study, 237 were screened; 226 were enrolled to open-label treatment epoch; 201 (88.9%) completed treatment epoch; 209 (92.5%) entered the post-treatment follow-up epoch and 152 (67.3%) completed the post-treatment follow-up epoch
Period: Overall Study
Arm/Group | Ligelizumab
Started | 226
Completed | 201
Not Completed | 25
Not completed — Adverse Event | 8
Not completed — Lack of Efficacy | 8
Not completed — Pregnancy | 3
Not completed — Protocol Violation | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The Safety set (SS) included all subjects who received at least one dose of study drug during this open-label study.
Arm/Group | Ligelizumab
Number analyzed (Participants) | 226
Age, Continuous [Mean (Standard Deviation); unit: years] — age
  years | 44.5 (12.69)
Age, Customized [Number; unit: participants]
  <65 years | 211
  >= 65 years | 15
Sex/Gender, Customized [Number; unit: Percentage of Participants] — Population: The Safety set (SS) included all subjects who received at least one dose of study drug during this open-label study.
  Percentage of Participants
    Female: number analyzed (Participants) | 170
    Female | 75.2
    Male: number analyzed (Participants) | 56
    Male | 24.8
Race/Ethnicity, Customized [Number; unit: Percentage of participants] — Population: The Safety set (SS) included all subjects who received at least one dose of study drug during this open-label study.
  Percentage of participants
    Asian: number analyzed (Participants) | 51
    Asian | 22.6
    Black or African American: number analyzed (Participants) | 3
    Black or African American | 1.3
    White: number analyzed (Participants) | 163
    White | 72.1
    American Indian or Alaska Native: number analyzed (Participants) | 1
    American Indian or Alaska Native | 0.4
    Unknown: number analyzed (Participants) | 2
    Unknown | 0.9
    Other: number analyzed (Participants) | 6
    Other | 2.7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment Emergent Adverse Event (AE)
Description: The primary objective of this study was to assess the long-term safety of one-year treatment of QGE031 in adult Chronic Spontaneous Urticaria (CSU) patients who completed the core study CQGE031C2201 using the following evaluations: number of participants with treatment emergent AEs of non-serious and serious nature including any events of special interest.
Time Frame: Within 16 weeks after Week 48
Population: Safety Set: All 226 subjects who received at least one dose of study drug during this open-label study were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab
Number analyzed (Participants) | 226
Participants | 190

2. Secondary Outcome: Percentage of Subjects Having Achieved UAS7 ≤ 6
Description: The secondary objective of this study was to assess the long-term efficacy of QGE031 in adult CSU patients who completed the CQGE031C2201 study using the following evaluations:
  Sustained remission defined as maintaining (Urticaria Activity Score) UAS7 ≤ 6 over 48 weeks post-treatment follow up epoch among the participants achieving remission at the end of treatment epoch.
Time Frame: Baseline, Week 52 and Week 100
Population: Safety Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ligelizumab
Number analyzed (Participants) | 226
percentage of participants
  Baseline | 0.44 [0 to 2.4]
  Week 52 | 61.06 [54.4 to 67.5]
  Week 100 | 28.32 [22.5 to 34.7]

3. Secondary Outcome: Number and Proportion of Participants Who Achieved UAS7≤ 6
Description: Summary of subjects with UAS7 ≤ 6. The long term efficacy of one-year treatment of ligelizumab 240 mg s.c. q4w is assessed by number and proportion of participants who achieved well controlled disease (UAS7≤ 6) at end of the treatment period (Week 52) and end of follow up period (Week 100).
Time Frame: Baseline, Week 52, Week 100
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab
Number analyzed (Participants) | 226
Participants
  Baseline | 1
  Week 52 | 138
  Week 100 | 64

ADVERSE EVENTS:
Time Frame: Within 16 weeks after Week 48
Description: Adverse Events (AEs) are any untoward sign or symptom that occurs during the study treatment
Groups:
- QGE031 240 mg q4w (TEAE): QGE031 240 mg every four weeks (TEAE)
- QGE031 240 mg q4w (Non-TEAE): QGE031 240 mg every four weeks (non-TEAE)
Arm/Group | QGE031 240 mg q4w (TEAE) | QGE031 240 mg q4w (Non-TEAE)
All-Cause Mortality (participants affected / at risk) | 1/226 | 0/226
Serious Adverse Events (participants affected / at risk) | 15/226 | 6/226
Other Adverse Events (participants affected / at risk) | 133/226 | 38/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QGE031 240 mg q4w (TEAE) (N=226) | QGE031 240 mg q4w (Non-TEAE) (N=226)
Angina pectoris (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Mouth cyst (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Complicated appendicitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QGE031 240 mg q4w (TEAE) (N=226) | QGE031 240 mg q4w (Non-TEAE) (N=226)
Injection site erythema (General disorders) | 13 | 0
Nasopharyngitis (Infections and infestations) | 57 | 10
Sinusitis (Infections and infestations) | 13 | 2
Upper respiratory tract infection (Infections and infestations) | 23 | 3
Urinary tract infection (Infections and infestations) | 12 | 3
Blood creatinine increased (Investigations) | 12 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 2
Headache (Nervous system disorders) | 29 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 23 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-10-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT02649218/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT02649218/SAP_001.pdf